CLINICAL TRIAL: NCT03264209
Title: Smart After-Care in Patients With Prostate Cancer: a Randomized Controlled Trial
Brief Title: Smart After-Care in Patients With Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ji Youl Lee (Other)
Responsible Party: Sponsor-Investigator, Ji Youl Lee, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KC17FNDI0557
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Case management (Experimental): Case management consists confirmation of hospital visit date, checking the efficacy of intervention, adverse effect and treatment compliance
  Interventions: Behavioral: Smart After-Care (Mobile health)
- Control: usual care (No Intervention): Usual care is provided with life style intervention including exercise and nutrition by printed materials.

INTERVENTIONS:
Behavioral: Smart After-Care (Mobile health) — Patients in intervention group will be provided with Smart After-Care Service including intervention for physical activity (aerobic exercise at least 90 or 150 minutes every week for 12 weeks depending on patients' aerobic fitness by monitoring with smartband and strengthening exercise at least 2 times a week for 12 weeks), information for prostate cancer and adequate life style, and smartband that can connect to the smartphone. Case management consists confirmation of hospital visit date, checking the adverse effect and treatment compliance.
  Arms: Intervention: Case management

SUMMARY:
This study aims to examine whether Smart After-Care service (Internet-and mobile-based lifestyle intervention) has an effect on patients' satisfaction and clinical outcomes in patients with prostate cancer on androgen deprivation therapy. Patients with prostate cancer on androgen deprivation therapy will participate in the study. The study design is a randomized controlled trial. The patients were randomly assigned to intervention or usual care groups. Intervention patients received Smart After-Care service for 3 months. Primary endpoint was an increase in patients' physical function as assessed using 2 minute walking test. Secondary endpoints included improvement in muscle strength, short physical performance battery, body composition, and health-related quality of life.

DETAILED DESCRIPTION:
After-care is a process targeted towards restoration or maintenance of the physical, mental, intellectual and social abilities of an individual affected by cancer. Internet-and mobile-based lifestyle intervention have emerged as potential modalities to complement and increase accessibility to after-care. In order to meet the growing need for after-care services, we developed a Smart after-care system that will assess the efficacy of a web-based smartphone-enabled intervention. The system provided specialized tools on after-care of prostate cancer including information on nutrition, physical activity, medication adherence, and mobile device that can connect to the smartphone. Patients with prostate cancer on androgen deprivation therapy will be screened for having adequate musculoskeletal and cardiopulmonary function.The study design is a randomized controlled trial. The patients were randomly assigned to intervention or usual care groups. Intervention patients received Smart After-Care management for 3 months. Primary endpoint was an increase in patients' physical function as assessed using 2 minute walking test. Secondary endpoints included improvement in muscle strength, short physical performance battery, body composition, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males diagnosed with prostate cancer
* Current treatment with ADT (GnRH agonist/antagonist with or without antiandrogen) for a minimum of 6 months after randomization
* Having Android smartphone

Exclusion Criteria:

* Having another (active) malignant disease within 3 month before randomization
* Having severe cardiopulmonary disease
* Having bone pain due to bone metastasis, (or) pathologic fracture
* Receiving total knee replacement arthroplasty, (or) total hip replacement arthroplasty
* No permission from treating/study physician to participate in exercise

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Physical function (2 minute walking test) | 3 months after randomization
  Cardiorespiratory endurance was examined by 2MWT performed on a 15.2-m hallway out-and-back course. Patients were instructed to walk as fast as they could until asked to stop at 2 min; the distance covered was recorded.

SECONDARY OUTCOMES:
Changes in muscle strength | 3 months after randomization
  A handgrip strength test was used to assess upper extremity muscle strength using a hand-held dynamometer. Patients were instructed to apply maximal power for 3 s with the shoulder adducted and neutrally rotated, elbow flexed at 90°, and the forearm and wrist in a neutral position. Three attempts were given with each hand and the best score (kg) for each was recorded. A 30-s chair stand test was used as a measure of lower extremity muscle strength. Each patient was seated in the middle of the chair (seat height of 40 cm, without armrests but with a backrest) with their back straight and both arms folded across their chest. The patients were instructed to stand up and sit down repetitively and encouraged to complete as many full stands as possible for 30 s while the instructor kept count.
Changes in short physical performance battery | 3 months after randomization
  The SPPB is calculated from three components: the ability to stand for up to 10 seconds with feet positioned in three ways (together side-by-side, semi-tandem and tandem); time to complete a 3-m or 4-m walk; and time to rise from a chair five times.
Changes in body composition | 3 months after randomization
  weight in kilograms, height in meters, body fat mass in kilograms, skeletal muscle mass in kilograms
Changes in health-related quality of life by EORTC QLQ-C30 | 3 months after randomization
  Units on a Scale
Changes in health-related quality of life by EORTC QLQ-PR25. | 3 months after randomization
  Units on a Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ji Youl Lee, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea